CLINICAL TRIAL: NCT06786273
Title: Time Course of Endometrium's Gene Expression and DNA Methylation Profiles Using Endometrial Tissue and Blood Samples
Brief Title: Time Course of Endometrium's Gene Expression Profiles Using Endometrial Tissue and Blood Samples
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Inti Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CS2-22033
Record Dates: First submitted 2025-01-15; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Fertility
Keywords: miRNAs; microRNAs; time course; blood

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- P+3 (Other): Women who get their blood drawn and endometrial tissue biopsy taken at 3 days after progesterone administration starts.
  Interventions: Genetic: Small RNA sequencing
- P+4 (Other): Women who get their blood drawn and endometrial tissue biopsy taken at 4 days after progesterone administration starts.
  Interventions: Genetic: Small RNA sequencing
- P+5 (Other): Women who get their blood drawn and endometrial tissue biopsy taken at 5 days after progesterone administration starts.
  Interventions: Genetic: Small RNA sequencing
- P+6 (Other): Women who get their blood drawn and endometrial tissue biopsy taken at 6 days after progesterone administration starts.
  Interventions: Genetic: Small RNA sequencing
- P+7 (Other): Women who get their blood drawn and endometrial tissue biopsy taken at 7 days after progesterone administration starts.
  Interventions: Genetic: Small RNA sequencing

INTERVENTIONS:
Genetic: Small RNA sequencing — The blood and endometrial tissue samples collected from the study groups will undergo small RNA sequencing to investigate the microRNA expression profiles associated with that phase.

SUMMARY:
This study aims to investigate whether the expression levels of microRNA (miRNA) in endometrial tissue and blood samples at various time points after ovulation can serve as biomarkers for assessing endometrial receptivity.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycle of 28-32 days.
* Between 25-38 years old.
* BMI between 18 to 30.
* Endogenous progesterone (P4) level of < 1 ng/mL prior to exogenous progesterone administration

Exclusion Criteria:

* Suspected intrauterine abnormality.
* Women who are breastfeeding
* Have a history of pelvic inflammatory disease, reproductive tract-related diseases, sexually transmitted diseases, systemic diseases or endocrine diseases.
* History of major illness.
* Use of hormonal contraceptives or intrauterine devices in the past 3 months.

Ages: 25 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 62 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
miRNA expression profiles | 1 month
  The samples collected would undergo small RNA sequencing in order to investigate the miRNA expression profiles of the patients and differences in expression profiles between the different intervention groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Lee Women's Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No